CLINICAL TRIAL: NCT02901990
Title: Observational Cohort Study to Evaluate Immunogenicity, Protection, and Persistence of Antibody to Mumps in 3-7 Years' Children Received One-dose Mumps-containing Vaccine
Brief Title: Observational Study to Assess Protection to Mumps in Children Received One-dose Mumps-containing Vaccine
Status: Completed | Type: Observational
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Other Study IDs: JSEPI001
Record Dates: First submitted 2016-09-02; First posted 2016-09-15 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Parotid Gland Infection; Fever
Keywords: mumps; immunity; cohort study; children; vaccine
MeSH Terms: conditions — Fever; Mumps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GMT-low-level group: low geometric mean titer (GMT) detected in the children who had received one-dose mumps-containing vaccine from precious cross sectional study
- GMT-high-level group: high geometric mean titer (GMT) detected in the children who had received one-dose mumps-containing vaccine from precious cross sectional study

SUMMARY:
This study was aimed to conduct a 3-year perspective study to observe the immunological effect of one-dose mumps-containing vaccine, monitor the incidence of mumps in vaccinated population aged 3-7 years，and provide basis for adjusting MMR immunization strategy in Jiangsu province, China.

DETAILED DESCRIPTION:
in 3-7 years old children with high risk of mumps, epidemiological investigation of the serum IgG antibody level were conducted, and then a prospective observational cohort was established in the population with a history of mumps vaccination, and the incidence of mumps in each antibody level group will be observed, the relationship between different antibody levels and the incidence after mumps vaccinated were analyzed, to explore attenuation of mumps IgG antibody levels in the body,S79 vaccine strain against F genotype mumps' antigenic cross-reactivity and the protective effect of antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3-7 years old;
2. local resident children living at least 3 months;
3. physical health, has been vaccinated at least once a dose of MuV

Exclusion Criteria:

1. did not administer MuV;
2. refused to collect venous blood;
3. have been infected with mumps;
4. have serious illness or other reasons should not participate in the study after clinical evaluation

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children aged 3-7 years who received as least one dose mumps-containing vaccine
Sampling Method: Probability Sample
Enrollment: 7901 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
to describe the sero-prevalence in specific age groups following an active surveillance of vaccinated subjects in each year | 3 years

SECONDARY OUTCOMES:
to describe wane immunity of IgG antibody to mumps virus in specific age groups following an active surveillance of vaccinated subjects in each year | 3 years
To characterize the incidence of mumps in specific age groups following an active surveillance of vaccinated subjects in each year | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Fenyang Tang, Principal Investigator — Jiangsu provincial CDC
Locations (6):
- China (6):
  - wujin district CDC, Changzhou, Jiangsu
  - lianshui county CDC, Huaian, Jiangsu
  - ganyu district CDC, Lianyungang, Jiangsu
  - gaogang district CDC, Taizhou, Jiangsu
  - tongshan district CDC, Xuzhou, Jiangsu
  - danyang county CDC, Zhenjiang, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun J, Li M, Zhang L, Deng X, Hu Y, Chen Q, Wang Z, Sun X, Liu Y. Mumps-specific antibody persistence in children aged 3-7 years immunized with two doses of mumps-containing vaccines: A prospective cohort study in Jiangsu Province, China. Hum Vaccin Immunother. 2023 Dec 31;19(1):2166758. doi: 10.1080/21645515.2023.2166758. Epub 2023 Jan 18. PMID 36653029
- [Derived] Liu Y, Liu Z, Deng X, Hu Y, Wang Z, Lu P, Guo H, Sun X, Xu Y, Tang F, Zhu FC. Waning immunity of one-dose measles-mumps-rubella vaccine to mumps in children from kindergarten to early school age: a prospective study. Expert Rev Vaccines. 2018 May;17(5):445-452. doi: 10.1080/14760584.2018.1445529. Epub 2018 Mar 12. PMID 29478347